CLINICAL TRIAL: NCT02042794
Title: Randomised Controlled Trial of Pringle Manoeuvre Versus Portal Vein Clamping in Patients Undergoing Liver Resection for Colorectal Liver Metastasis - A Pilot Study
Brief Title: Pringle Manoeuvre Versus Portal Vein Clamping for Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PB-PG-0711-25080
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Liver Metastasis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Liver resection is an operation to remove the diseased part of the liver. The liver is supplied by two vessels, the hepatic artery and the portal vein supplying 25% and 75% respectively of the total blood flow with 50% oxygen from each vessel. During liver resection it is standard practice to clamp both vessels(Pringle's manoeuvre), so as to avoid bleeding. Clamping both the vessels deprives the unaffected liver from nutrients required for survival. Reinstating the blood supply causes further damage by pouring harmful substances into the liver, which accumulate during the clamping. We hypothesize that not clamping the oxygen rich hepatic artery will cause less damage to the liver.

Our aim is to compare the Pringle manoeuvre with portal vein clamping, to identify if the latter will result in less tissue injury and thereby fewer complications. Initially we aim to conduct a pilot study. The main objective is to ensure that patients can be successfully recruited and that data capture is complete. The secondary outcomes will be development of infective complications by 30 days following surgery, bleeding and blood transfusion requirements, heart/chest complications, recovery of liver functions, growth of remnant liver, death within 30 days following surgery, length of high dependency unit/hospital stay and quality of life at 3 months after surgery.

There is published literature on the safety of this method and in the event of any intraoperative problems, the procedure will be converted to the standard Pringle manoeuvre. The Liver Unit at St James's University Hospital has four surgeons performing around 270 liver cancer resections per year, of which nearly 160 are for bowel cancer spread. Considering the team's experience in research and liver surgery, we believe it is well placed to conduct the trial in a safe and efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing liver resection for CRLM
* Portal venous clamping as considered appropriate
* Participating patients should be able to understand the study objectives and be able to give written consent
* Able to complete study questionnaire

Exclusion Criteria:

* Patients having simultaneous bowel and hepatic surgery
* Patients participating in other trials that could impact the outcomes measures being recorded
* Patients who are pregnant
* Patients taking immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer, inflammatory and immune study, oral and gastrointestinal.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The ability to recruit and randomise patients into the study | 14months

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom